CLINICAL TRIAL: NCT02530775
Title: "Is Instrumentation Necessary for "Static" Degenerative Spondylolisthesis - A Prospective Randomized Clinical Study"
Brief Title: "Is Instrumentation Necessary for "Static" Degenerative Spondylolisthesis"
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not receive IRB approval and was withdrawn
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Joon Yung Lee, MD, M.D., University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO15040227
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Degenerative Spondylolisthesis; Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- instrumented arthrodesis (Active Comparator): Degenerative Spondylolisthesis and Spinal Stenosis patients having a surgical procedure. The surgical procedure is the intervention and is a spinal fusion with use of instrumentation and lumbar laminectomy. No additional "drug" or "device" intervention.
  Interventions: Procedure: instrumented spinal fusion with laminectomy
- non-instrumented arthrodesis (Active Comparator): Degenerative Spondylolisthesis and Spinal Stenosis patients having a surgical procedure. The surgical procedure is the intervention and is a spinal fusion without the use of instrumentation and lumbar laminectomy. No additional "drug" or "device" intervention.
  Interventions: Procedure: non-instrumented spinal fusion with laminectomy

INTERVENTIONS:
Procedure: instrumented spinal fusion with laminectomy — Once determined that a patient has single level "static" degenerative spondylolisthesis and is planning to schedule surgery the patient will be approached by a research team member explaining the study and reviewing the informed consent document. If the patient chooses to participate, he or she will be randomized to be apart of the non-instrumented arthrodesis with laminectomy group or the instrumented arthrodesis with laminectomy group. Both are standard approved surgical approaches; however, using instrumentation is the more commonly used approach.
  Arms: instrumented arthrodesis
Procedure: non-instrumented spinal fusion with laminectomy — Once determined that a patient has single level "static" degenerative spondylolisthesis and is planning to schedule surgery the patient will be approached by a research team member explaining the study and reviewing the informed consent document. If the patient chooses to participate, he or she will be randomized to be apart of the non-instrumented arthrodesis with laminectomy group or the instrumented arthrodesis with laminectomy group. Both are standard approved surgical approaches; however, using instrumentation is the more commonly used approach.
  Arms: non-instrumented arthrodesis

SUMMARY:
The purpose of this study is to determine whether instrumented lumbar fusion provides superior clinical outcomes in comparison to non-instrumented fusion in patients with "static" degenerative spondylolisthesis.

DETAILED DESCRIPTION:
This study will determine whether instrumented lumbar fusion will provide superior clinical outcomes in comparison to non-instrumented fusion in patients with "STATIC" degenerative spondylolisthesis. At the time of scheduling surgery, patients who meet the inclusion/exclusion criteria will be asked to participate. Patients who agree, will be randomized to either non-instrumented or instrumented arthrodesis group. Intra-operative, peri-operative, and post-operative data will be collected and compared. The investigators predict to get very similar clinical outcomes between the two groups, with possibly less complications from the non-instrumented group and definitely a reduction in cost compared to the instrumented group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable L4-5 spondylolisthesis on lumbar flexion and extension radiographs. Stability will be determined by the treating physician.
2. Patients with concomitant spinal stenosis.
3. Laminectomy at any lumbar levels of stenosis.
4. Fusion only at L4-5 level.

Exclusion Criteria:

1. Prior lumbar spine surgery
2. Multi-level spondylolisthesis
3. Anterior interbody work/fusion
4. Tumor
5. Infection
6. Trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional Outcome Scores: SF-12/SF-36 Quality of Life Questionnaires | Up to 2 years
  Measured by patient outcome survey such as the SF-12 or SF-36 Questionnaire (all questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible)
Functional Outcome Scores: Oswestry Disability Index (ODI) Questionnaire | Up to 2 years
  Measured by patient outcome survey such as the Oswestry Disability Index (ODI) that assesses low back pain (scoring ranges from 0 to >35)

SECONDARY OUTCOMES:
Rate of Infection | Expected average of 4 weeks
  Wound Complications
Rate of Symptomatic Pseudoarthrosis | Up to 2 years
Need for Revision Surgery | Up to 2 years
  Return to the OR
Length of Hospital Stay | Expected average of 1 week
Surgical Time | 2-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joon Y Lee, M.D., Principal Investigator — University of Pittsburgh Medical Center